CLINICAL TRIAL: NCT06369974
Title: An Open-label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for TUBB4A-related Leukodystrophy
Brief Title: Single Participant Study of an Experimental ASO Treatment for TUBB4A-related Leukodystrophy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: n-Lorem Foundation (Other)
Responsible Party: Principal Investigator, Florian Eichler, Director of the Center for Rare Neurological Diseases, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000386
Record Dates: First submitted 2024-03-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Genetic Disease
Keywords: leukodystrophy; antisense oligonucleotide; TUBB4A-related leukodystrophy; Hypomyelination; ASO
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Single participant interventional study
Masking Description: Open label study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Open Label
  Interventions: Drug: Antisense oligonucleotide treatment (ASO)

INTERVENTIONS:
Drug: Antisense oligonucleotide treatment (ASO) — Drug: nL-TUBB4-001; Personalized antisense oligonucleotide
  Other Names: nL-TUBB4-001

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single pediatric participant with TUBB4A associated leukodystrophy.

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single pediatric participant with a de novo pathogenic gain of function TUBB4A mutation associated with severe leukodystrophy with hypomyelination with atrophy of the basal ganglia and cerebellum (H-ABC)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Clinical phenotype and neuroimaging consistent with a diagnosis of TUBB4A-related leukodystrophy/Hypomyelination with Atrophy of the Basal Ganglia and Cerebellum (H-ABC)
* Documented genetic mutation in TUBB4A

Exclusion Criteria:

* Participant has any known contraindication to or unwillingness to undergo lumbar puncture
* Use of investigational medication within 5 half-lives of the drug at enrolment
* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Neurological assessments | Baseline to 24 months
  Change from baseline at 24 months post nL-TUBB4-001 administration in scores on the GMFM88, HINE-1, HINE-2, Bayley-4, and Vineland-3 developmental assessment scales, as well as the Tardieu Spasticity Scale and PedsQL Family Impact Module

SECONDARY OUTCOMES:
Feeding and swallow evaluation | Baseline to 24 months
  Change from baseline at 24 months post nL-TUBB4-001 administration in assessment of feeding and swallow evaluation.
Safety and tolerability | Baseline to 24 months
  Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Florian Eichler, MD, Principal Investigator — Massachusetts General Hospital